CLINICAL TRIAL: NCT05139654
Title: Shoulder Kinematics and Muscle Activation in Sport Climbers With Shoulder Pain
Status: Completed | Type: Observational
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Yin-Liang Lin, Assistant Professor, National Yang Ming Chiao Tung University
Other Study IDs: YM110156E
Record Dates: First submitted 2021-11-17; First posted 2021-12-01 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: Shoulder Pain; Shoulder Impingement Syndrome
Keywords: Sport climbing; Shoulder kinematics; Electromyography; Shoulder pain
MeSH Terms: conditions — Shoulder Pain; Shoulder Impingement Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Shoulder pain climbers group: Subjects with shoulder pain will be included to perform scaption and pull-up, and assess shoulder kinematics and muscle activation at the same time.
  Interventions: Other: Arm elevation in the scapular plane; Other: Pull up with gymbar; Other: Pull up with fingerboard
- Healthy climbers group: Healthy subjects will be included to compare the differences in shoulder kinematics and muscle activation between healthy subjects and subjects with shoulder pain. Subjects in this group will received the same assessments as the shoulder pain climbers group.
  Interventions: Other: Arm elevation in the scapular plane; Other: Pull up with gymbar; Other: Pull up with fingerboard

INTERVENTIONS:
Other: Arm elevation in the scapular plane — Lift the arm up in the scapular plane
Other: Pull up with gymbar — Grasp the gymbar with both hands and pull up as high as the subject can
Other: Pull up with fingerboard — The width of the fingerboar is 20 mm. Pull up with fingers on the fingerboard.

SUMMARY:
Sport climbing has recently become a highly popular sport and was included in the Summer Olympic Games 2021. Shoulder injury accounts for 15 to 20 percent of all sport climbing injuries, and it is the third most common problems, only surpassed by wrist and hand injuries. Sport climbing involves both open and closed chain movements of upper limbs. These prolonged and repetitive movements on vertical or overhanging terrain may lead to overuse and fatigue, which result in injuries. Sport climbing consists of multiple movement elements. Pull up with small holds is a basic movement in sport climbing, and activates many shoulder muscles, including trapezius, serratus anterior, latissimus dorsi. Studies related to sport climbing have focused on observing difference between sport climbers and non-sport climbers. Altered posture, increased scapulohumeral rhythm during arm elevation, and decreased shoulder angle during one-arm hanging have been observed in sport climbers. However, little studies have investigated whether climbers with shoulder injuries demonstrate different shoulder kinematics and muscle activation during tasks related to sport climbing. Therefore, the purpose of this study is to investigate the shoulder kinematics and muscle activation during pull-up with small holds in sport climbers with and without shoulder pain. Methods. Thirty sport climbers with shoulder pain and 30 healthy control subjects matched with gender, age, dominant hand and experience will be recruited in this study. All subjects will undertake physical examinations such as shoulder range of motion (ROM). Shoulder kinematics and muscle activation will be collected during arm elevation in the scapular plane and pull-up with gym-bar and 20mm depth small climbing holds. An electromagnetic tracking system will be used to measure bilateral scapular and humerothoracic kinematics. Surface electromyography (EMG) will be used to record muscle activation of bilateral upper trapezius, lower trapezius, serratus anterior and latissimus dorsi. Demographic data and physical examination will be analyzed by independent t test or Chi-square test. Two-way ANOVA will be used to test differences between groups in kinematics and EMG data at different phases of tasks. If significant interaction effect is found, Post-hoc pairwise comparison with Bonferroni correction will be used. The significant level is set at 0.05.

ELIGIBILITY:
Inclusion Criteria of Patients with Shoulder Pain:

1. Ages ranges from 20-40 years old
2. At least one year of experience of sport climbing
3. Sport Climbing frequency ≥ 6 hours per week in the last one month
4. Shoulder pain ≥ 1 month
5. Minimum of 3/10 on the numerical rating scale (NRS) in the last one month

Inclusion Criteria of Healthy Subjects in the control group:

1. Ages ranges from 20-40 years old
2. Gender, age, dominant hand and experience matching to shoulder pain climbers group
3. At least one year of experience of sport climbing
4. Sport Climbing at least 6 hours per week in the last one month
5. No history of shoulder pain in the last six months

Exclusion Criteria of Patients with Shoulder Pain and All Healthy Subjects

1. History of upper limb surgery or fracture
2. History of shoulder dislocation
3. History of neck pain, back pain, or elbow injuries in the last one year
4. Wrist or finger pain during sport climbing > 3/10 on the numerical rating scale (NRS)
5. Shoulder pain during pull-up > shoulder pain during sport climbing
6. Intensive exercise within 12 hours or any delay onset muscle soreness
7. Systemic autoimmune disease
8. Cancer
9. Pregnancy

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 1. Ages ranges from 20-40 years old
  2. At least one year of experience of sport climbing
  3. Sport Climbing frequency ≥ 6 hours per week in the last one month
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-11-10 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2022-06-10 (Actual)

PRIMARY OUTCOMES:
Shoulder kinematics during arm elevation | Immediately during the experiment
  Scapular kinematics, including anterior/posterior tilt, upward/downward rotation, and internal/external rotation in scapular plane elevation at 30°, 60°, 90°, and 120°, and will be described with degree (°).
Shoulder kinematics during pull-up with gym-bar | Immediately during the experiment
  Scapular kinematics, including anterior/posterior tilt, upward/downward rotation, and internal/external rotation in pull-up, and will be described with degree (°).
Shoulder kinematics during pull-up with finger board | Immediately during the experiment
  Scapular kinematics, including anterior/posterior tilt, upward/downward rotation, and internal/external rotation in pull-up, and will be described with degree (°).
Scapular muscles activation during arm elevation | Immediately during the experiment
  The root mean square of electromyography (EMG) data of the upper trapezius, lower trapezius, serratus anterior, and latissimus dorsi will be normalized by the maximum voluntary contraction amplitude (percentage of maximal voluntary contraction, %) and calculated over three 30° increments of motion during arm elevation from 30° to 120°, including 30° - 60°, 60° - 90°, and 90° - 120°.
Scapular muscles activation during pull-up with gym-bar | Immediately during the experiment
  The root mean square of electromyography (EMG) data of the upper trapezius, lower trapezius, serratus anterior, and latissimus dorsi will be normalized by the maximum voluntary contraction amplitude (percentage of maximal voluntary contraction, %).
Scapular muscles activation during pull-up with finger board | Immediately during the experiment
  The root mean square of electromyography (EMG) data of the upper trapezius, lower trapezius, serratus anterior, and latissimus dorsi will be normalized by the maximum voluntary contraction amplitude (percentage of maximal voluntary contraction, %).

CONTACTS AND LOCATIONS:
Overall Officials: Yin-Liang Lin, Principal Investigator — National Yang Ming Chiao Tung University
Locations (1):
- National Yang Ming University, Taipei, Taiwan